CLINICAL TRIAL: NCT03131960
Title: A Pivotal Randomized Study Assessing Vagus Nerve Stimulation (VNS) During Rehabilitation for Improved Upper Limb Motor Function After Stroke (VNS-REHAB)
Brief Title: Pivotal Study of VNS During Rehab After Stroke (VNS-REHAB)
Acronym: VNS-REHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroTransponder Inc. (Industry)
Collaborators: ResearchPoint Global (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-St-03
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cerebrovascular Stroke; Upper Extremity Paresis
MeSH Terms: conditions — Stroke; Paresis | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, parallel study with partial crossover (control subjects crossover to treatment after randomized portion)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, therapists (care providers), investigators, and outcomes assessors do not know which group (VNS or control VNS) the patients are randomized. Only one person at the site - the programmer who programs the device settings - knows which group the subject is randomized into.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- VNS + Rehabilitation (1) (Experimental): Study treatment is vagus nerve stimulation (VNS) delivered during rehabilitation.
  Interventions: Device: Paired Vagus Nerve Stimulation; Other: Rehabilitation
- Control VNS (Active Comparator): Active control treatment is rehabilitation (standard-of-care treatment) with only a minimal amount of VNS at the start of each session intended to support blinding.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Device: Paired Vagus Nerve Stimulation — Stimulation of the vagus nerve that is paired with upper limb rehabilitation movements.
  Arms: VNS + Rehabilitation (1)
Other: Rehabilitation — Rehabilitation movements to improve upper limb function after stroke

SUMMARY:
This is a pivotal phase study of up to 120 subjects and 15 clinical sites. All subjects are implanted with the Vivistim System® and then randomized to either study treatment or active-control treatment. The randomization will be stratified by age (<30, >30) and baseline FMA UE (20 to <35; >35 to 50). Study treatment is vagus nerve stimulation (VNS) delivered during rehabilitation. Active control treatment is rehabilitation (standard-of-care treatment) with only a minimal amount of VNS at the start of each session intended to support blinding.

DETAILED DESCRIPTION:
This study has three distinct stages: Stage I, an acute blinded stage, Stage II, an unblinded stage through one year of standard VNS, and Stage III, an unblinded stage for yearly follow-up after one year of VNS. The Control group crosses over to VNS treatment at Stage II.

For Stage I, subjects have:

* consent and evaluation (screening),
* one pre-implant evaluation,
* surgical implant of the device system and randomization into one of the treatment arms,
* one baseline evaluation after device implant surgery but before initiation of treatment,
* 6 weeks of treatment (standard-of-care rehabilitation + standard VNS or standard-of-care rehabilitation + active control VNS), and then
* post-acute therapy evaluations at 1, 30 and 90 days after the 6 weeks of treatment.
* Between Day 1 (V5) and Day 30 (V6) post-acute therapy, both groups will receive in-home, self-directed rehabilitation (30 minutes of daily rehabilitation as assigned by the therapist) with either in-home activated VNS (VNS group) or no VNS (Control group). This means that the control subjects will not have the in-home activated VNS until they complete the second 6-week session of in-clinic rehabilitation with follow-up assessments as described below in Stage II. At this point (Day 30) subjects start scheduling for their continuing long-term follow-up.
* Between Day 30 and Day 90 post-acute therapy, both groups continue in-home, self-directed rehabilitation (30 minutes of daily rehabilitation as assigned by the therapist). The VNS group continues to receive in-home VNS with magnet use; the Control group continues to use the magnet but does not receive any VNS. The Day 90 post-acute therapy visit is V7; it is the first quarterly visit (3 months after study therapy) for the VNS group and is the re-baseline visit (visit just prior to the initiation of standard VNS therapy) for the Control group.

Stage II:

* VNS subjects will continue to have quarterly assessments through the end of the first year (6m, 9m, 12m).
* Subjects in the control group will crossover for a second 6-week in-clinic rehabilitation period where they will now receive rehabilitation with standard VNS.
* Control subjects will then have the three post therapy assessments (1, 30 and 90 days after therapy ends); in-home VNS initiated by a magnet swipe starts at the Post-1 visit (LT1). Thereafter, control subjects will follow the same schedule as VNS subjects for the remainder of the study (6m, 9m, 12m follow-ups, plus yearly visits thereafter).
* Subjects in both groups will receive "booster" in-clinic rehabilitation plus VNS therapy sessions one month prior to their 6- and 12-month assessment visits. These sessions occur on three days over a one-week period (typically Mon, Wed, Fri).

Stage III:

• After one year of standard VNS therapy (~13.5 months after implant for VNS group subjects and ~18 months after implant for Control group subjects), subjects who wish to keep their device for further use will have annual follow-up assessments until commercial approval.

ELIGIBILITY:
Inclusion Criteria:

1. History of unilateral supratentorial ischemic stroke that occurred at least 9 months but not more than ten 10 years prior to enrollment.
2. Age >22 years and <80 years.
3. FMA-UE score of 20 to 50 (inclusive of 20 and 50).
4. Ability to communicate, understand, and give appropriate consent. Subjects should be able to follow two-step commands.
5. Right- or left-sided weakness of upper extremity.
6. Active wrist flexion/extension; active abduction/extension of thumb and at least two additional digits.

Exclusion Criteria:

1. History of hemorrhagic stroke
2. Presence of ongoing dysphagia or aspiration difficulties.
3. Subject receiving medication that may significantly interfere with the actions of VNS on neurotransmitter systems at study entry. A list of excluded medications will be provided to Investigators.
4. Prior injury to vagus nerve, either bilateral or unilateral (e.g., injury during carotid endarterectomy).
5. Severe or worse depression (Beck Depression Scale > 29) (Beck et al., 1961)
6. Unfavorable candidacy for device implant surgery (e.g., history of adverse reactions to anesthetics, poor surgical candidate in surgeon's opinion, etc.)
7. Current use of any other stimulation device, such as a pacemaker or other neurostimulator; current use of any other investigational device or drug.
8. Medical or mental instability (diagnosis of personality disorder, psychosis, or substance abuse) that would prevent subject from meeting protocol timeline.
9. Pregnancy or plans to become pregnant or to breastfeed during the study period.
10. Current requirement, or likely future requirement, of diathermy during the study duration.
11. Active rehabilitation within 4 weeks prior to consent.
12. Botox injections or any other non-study active rehabilitation of the upper extremity within 4 weeks prior to therapy through the post-30 day visit (Visit 6).
13. Severe spasticity of the upper limb (Modified Ashworth ≥3) (Bohannon and Smith, 1987).
14. Significant sensory loss. Sensory loss will be measured using the Upper Extremity sensory section of the Fugl Meyer Assessment of Physical Performance. The assessment addresses light touch (2 items) and proprioception (4 items).The highest points attained is 12; subjects with scores less than 6 will be excluded from the study.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (15):
  - Perseverance Research Center, Scottsdale, Arizona
  - Rancho Research Institute, Downey, California
  - Providence St. John's Medical Center, Santa Monica, California
  - Mayo Jacksonville / Brooks Rehabilitation, Jacksonville, Florida
  - Emory University Medical School, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - New York Presbyterian Hospital / Weill Cornell Medicine, New York, New York
  - Burke Medical Research Institute, White Plains, New York
  - Ohio State University - Neuroscience Research Institute, Columbus, Ohio
  - Thomas Jefferson, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - TIRR Memorial Hermann (UT Health Science Center at Houston), Houston, Texas
- United Kingdom (5):
  - Royal Aberdeen Infirmary, Aberdeen
  - University of Glasgow, Queen Elizabeth University Hospital, Glasgow
  - Royal London, London
  - Newcastle (Royal Victoria Infirmary), Newcastle upon Tyne
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kimberley TJ, Prudente CN, Engineer ND, Pierce D, Tarver B, Cramer SC, Dickie DA, Dawson J. Study protocol for a pivotal randomised study assessing vagus nerve stimulation during rehabilitation for improved upper limb motor function after stroke. Eur Stroke J. 2019 Dec;4(4):363-377. doi: 10.1177/2396987319855306. Epub 2019 Jun 17. PMID 31903435
- [Background] Khodaparast N, Hays SA, Sloan AM, Fayyaz T, Hulsey DR, Rennaker RL 2nd, Kilgard MP. Vagus nerve stimulation delivered during motor rehabilitation improves recovery in a rat model of stroke. Neurorehabil Neural Repair. 2014 Sep;28(7):698-706. doi: 10.1177/1545968314521006. Epub 2014 Feb 18. PMID 24553102
- [Background] Dawson J, Pierce D, Dixit A, Kimberley TJ, Robertson M, Tarver B, Hilmi O, McLean J, Forbes K, Kilgard MP, Rennaker RL, Cramer SC, Walters M, Engineer N. Safety, Feasibility, and Efficacy of Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Ischemic Stroke. Stroke. 2016 Jan;47(1):143-50. doi: 10.1161/STROKEAHA.115.010477. Epub 2015 Dec 8. PMID 26645257
- [Result] Dawson J, Liu CY, Francisco GE, Cramer SC, Wolf SL, Dixit A, Alexander J, Ali R, Brown BL, Feng W, DeMark L, Hochberg LR, Kautz SA, Majid A, O'Dell MW, Pierce D, Prudente CN, Redgrave J, Turner DL, Engineer ND, Kimberley TJ. Vagus nerve stimulation paired with rehabilitation for upper limb motor function after ischaemic stroke (VNS-REHAB): a randomised, blinded, pivotal, device trial. Lancet. 2021 Apr 24;397(10284):1545-1553. doi: 10.1016/S0140-6736(21)00475-X. PMID 33894832
- [Derived] Kimberley TJ, Cramer SC, Wolf SL, Liu C, Gochyyev P, Dawson J; VNS-REHAB Trial Group. Long-Term Outcomes of Vagus Nerve Stimulation Paired With Upper Extremity Rehabilitation After Stroke. Stroke. 2025 Aug;56(8):2255-2265. doi: 10.1161/STROKEAHA.124.050479. Epub 2025 May 7. PMID 40329913
- [Derived] Lin S, Rodriguez CO, Wolf SL. Vagus Nerve Stimulation Paired With Upper Extremity Rehabilitation for Chronic Ischemic Stroke: Contribution of Dosage Parameters. Neurorehabil Neural Repair. 2024 Aug;38(8):607-615. doi: 10.1177/15459683241258769. Epub 2024 Jun 5. PMID 38836606
- [Derived] Vora I, Gochyyev P, Engineer N, Wolf SL, Kimberley TJ. Distal Versus Proximal Arm Improvement After Paired Vagus Nerve Stimulation Therapy After Chronic Stroke. Arch Phys Med Rehabil. 2024 Sep;105(9):1709-1717. doi: 10.1016/j.apmr.2024.05.018. Epub 2024 May 28. PMID 38815953
- See also: Study recruiting website — http://www.vnsstroketrial.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VNS + Rehabilitation (1) | Control VNS
Started | 53 (1 participant missed the day one visit (V5) but remained in the study and returned for the day 90 assessment (V7).) | 55 (1 discontinued treatment due to adverse event and inability to tolerate rehabilitation.)
Completed | 53 | 54
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VNS + Rehabilitation (1) | Control VNS | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 35 | 65
  >=65 years | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.2) | 61.1 (9.2) | 60.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 34 | 36 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 42 | 42 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 36 | 38 | 74
  United Kingdom | 17 | 17 | 34
FMA-UE Baseline Score [Mean (Standard Deviation); unit: units on a scale] — The upper extremity portion of the Fugl-Meyer Assessment (FMA-UE) was collected at each visit. The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment). The study allowed entry on the FMA-UE between 20 and 50.
  units on a scale | 34.4 (8.2) | 35.7 (7.8) | 35.1 (8.0)
WMFT Baseline Score [Mean (Standard Deviation); unit: units on a scale] — The Wolf Motor Function Test (WMFT) is an assessment scale of upper extremity functional level after stroke. The functional assessment range is an average of 15 sub-items with a range from 0 to 5, with 0 (meaning did not attempt) to 5 (meaning normal).
  units on a scale | 2.71 (0.70) | 2.83 (0.65) | 2.76 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment, Upper Limb (FMA-UE) Average Change
Description: The Fugl-Meyer Assessment, Upper Limb (FMA-UE) was analyzed for difference in average change at 1-day after 6-weeks of therapy compared to baseline (Difference in average change in FM-A from baseline [V4] to one day after therapy [V5]). The upper extremity portion of the Fugl-Meyer Assessment (FMA-UE) was collected at each visit. The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment).
Time Frame: V5, One day after 6-weeks of therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VNS + Rehabilitation (1) | Control VNS
Number analyzed (Participants) | 53 | 55
units on a scale | 5.0 (4.4) | 2.4 (3.8)
Statistical Analysis 1: Comparison: VNS + Rehabilitation (1) vs Control VNS; Test type: Superiority; p = 0.0014, ANCOVA

2. Secondary Outcome: Fugl-Meyer Assessment, Upper Limb (FMA-UE) Average Change
Description: The Fugl-Meyer Assessment, Upper Limb (FMA-UE) was analyzed for change in average score at 90-days after 6-weeks of therapy (change in average FMA-UE from baseline [V4] to 90 days after therapy [V7]). The upper extremity portion of the Fugl-Meyer Assessment (FMA-UE) was collected at each visit. The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment).
Time Frame: V7, 90 days after 6-weeks of therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VNS + Rehabilitation (1) | Control VNS
Number analyzed (Participants) | 53 | 55
units on a scale | 5.8 (6.0) | 2.8 (5.2)
Statistical Analysis 1: Comparison: VNS + Rehabilitation (1) vs Control VNS; ANCOVA; Test type: Superiority; p = 0.0077, ANCOVA

3. Secondary Outcome: Fugl-Meyer Assessment, Upper Limb (FMA-UE) Response
Description: The Fugl-Meyer Assessment, Upper Limb (FMA-UE) Response is the percent of patients with a 6 point or greater improvement on the (FMA-UE). The percent of patients with the 6-point change is calculated at 90-days after 6-weeks of therapy compared to baseline (V4). The upper extremity portion of the Fugl-Meyer Assessment (FMA-UE) was collected at each visit. The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment).
Time Frame: V7, 90 days after 6-weeks of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | VNS + Rehabilitation (1) | Control VNS
Number analyzed (Participants) | 53 | 55
Participants | 25 | 13
Statistical Analysis 1: Comparison: VNS + Rehabilitation (1) vs Control VNS; Test type: Superiority; p = 0.0098, Regression, Logistic

4. Secondary Outcome: Wolf Motor Function Test (WMFT) Average Change
Description: The Wolf Motor Function Test (WMFT) is an assessment scale of upper extremity functional level after stroke. The functional assessment range is an average of 15 sub-items with a range from 0 to 5, with 0 (meaning did not attempt) to 5 (meaning normal). WMFT 90-day - is a measure of the functional assessment change from baseline to 90 days after 6-weeks of therapy.
Time Frame: V7, 90 days after 6-weeks of therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VNS + Rehabilitation (1) | Control VNS
Number analyzed (Participants) | 53 | 55
units on a scale | 0.46 (0.40) | 0.16 (0.30)
Statistical Analysis 1: Comparison: VNS + Rehabilitation (1) vs Control VNS; Test type: Superiority; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of the randomized study (enrollment, 4-week baseline, implant, 2-week recover, 6-week therapy, 90-day follow-up) and reported here.
Arm/Group | VNS + Rehabilitation (1) | Control VNS
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/55
Serious Adverse Events (participants affected / at risk) | 5/53 | 3/55
Other Adverse Events (participants affected / at risk) | 43/53 | 42/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS + Rehabilitation (1) (N=53) | Control VNS (N=55)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — Patient with history of seizures had one during the 5th week of study treatment. Admitted to the ICU, recovered, was discharged, and continued in the study. The device implant and device stimulation are not related to this event (patient history).
Acute Kidney Injury (AKI)/ chronic kidney disease (CKD) (Renal and urinary disorders) | 0 (0) | 1 (1) — The patient was hospitalized after 7-8 months of worsening swelling and dyspnea on exertion (pre study). Found to have acute onset kidney injury (AKI on Chronic Kidney Disease [CKD]). Patient recovered and continued. Not related to implant or stim.
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 1 (1) | 0 (0) — Subject hospitalized with urinary tract infection. Subject recovered and continued in the study. No relationship to implant surgery or stimulation.
Dysphonia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Subject experienced vocal cord paresis and dysphonia after surgery. Recovered over 5 weeks; laryngoscope confirmed complete recovery. Related to the implant procedure but not stimulation. Subject recovered and continued in the study.
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) — 1 Subject fell at home walking down steps; fractured two vertebrae. 1 Subject fell at hospital during testing. 1 subject fell at home and broke her humerus. Subjects missed visits but continued in the study. No relationship to surgery or therapy.
Colinic Diverticular Abscess (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject reported pain and achiness at home. ER assessment indicated CDA. CDA drained and antibiotics started; subject returned home and recovered. No relationship to device implant or stimulation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS + Rehabilitation (1) (N=53) | Control VNS (N=55)
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (7)
Pain (General disorders) | 5 (5) | 7 (7)
Coughing/Hoarseness (Injury, poisoning and procedural complications) | 8 (8) | 10 (10)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3)
Low Mood (Psychiatric disorders) | 5 (5) | 4 (4)
Bruise (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2)
Local Throat Irritation (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Headache (Vascular disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT03131960/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT03131960/SAP_001.pdf